CLINICAL TRIAL: NCT02225691
Title: Effect of Introducing Daily Paired Testing to Poorly Controlled Chinese Diabetes Patients on Glycemic Control and Self Care
Brief Title: Effect of Paired Testing to Poorly Controlled Chinese Diabetes on Glycemic Control and Self Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai 6th People's Hospital (Other)
Responsible Party: Principal Investigator, Weiping Jia, The director of the endocrinology and metabolism department of the Shanghai 6th People's Hospital, Shanghai 6th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014-32
Record Dates: First submitted 2014-08-22; First posted 2014-08-26 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-11

CONDITIONS: Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1
Keywords: type 1 diabetes; type 2 diabetes; paired testing
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- paired testing of blood glucose (Experimental): Patient will be randomly assigned to one of 2 arms, namely (i) paired testing (PT) arm; and (ii) control (CL) arm. Paired testing arm will undergo paired testing of blood glucose.
  Interventions: Device: Paired testing of blood glucose Accu-Chek®
- control arm (No Intervention): Non-insulin patients will be randomly assigned to one of 2 arms, namely (i) paired testing (PT) arm; and (ii) control (CL) arm. Patients in the control arms will not undergo paired testing and will be managed as before.

INTERVENTIONS:
Device: Paired testing of blood glucose Accu-Chek® — Patients in the paired testing arms will undergo training on paired testing with Accu-Chek® Active blood glucose meters. The paired testing training would include (1) how and when (testing regimen) to perform paired testing, and (2) how to respond to paired testing readings via lifestyle modifications, self-adjustment of insulin dose and additional testing, if applicable. Please refer to Annex A for further details of the training.
  Other Names: Accu-Chek® Active blood glucose meters
  Arms: paired testing of blood glucose

SUMMARY:
This study aims is to evaluate the effect of introducing paired testing on actual testing frequency, glycemic control, psychosocial and behavioural aspects of poorly controlled diabetes patients in China.

DETAILED DESCRIPTION:
Self monitoring of blood glucose (SMBG) in insulin treated type 1 and type 2 diabetics has consistently been demonstrated to confer benefits, and is considered an essential part in the management of diabetes. In China, utilization of SMBG among diabetes patients is low. Even among those who perform SMBG regularly, the daily testing frequency falls short of those recommended in international and national clinical guidelines. There is thus a need to create the awareness of the benefits of SMBG and at the same time establish a SMBG regimen that is deemed practically feasible and cost effective for diabetes patients.

Paired testing entails the act of measuring glucose level before and after an event that may impact the glucose level in a patient, e.g. meals, exercise, medication adjustment, and thereafter responding to any abnormal glucose levels/patterns by modifying lifestyle and/or medication.

This study aims is to evaluate the effect of introducing paired testing on actual testing frequency, glycemic control, psychosocial and behavioral aspects of poorly controlled diabetes patients in China.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with diabetes mellitus
* HbA1c ≥ 8% measured within the a month prior to enrolment
* Have not been performing SMBG on a regular (daily) basis within the 3 months prior to enrolment
* Willing and able to use Accu-Chek® Active blood glucose meter to perform daily SMBG
* Willing and able to complete participant questionnaires
* Willing and able to visit the physician at month 3 and month 6
* Provide informed consent prior to enrolling in the study

Exclusion Criteria:

* Any retinopathy that required photocoagulation or retinal surgery in the 6 months prior to enrolment or that may require photocoagulation or retinal surgery during the study
* Any clinically significant condition that required hospitalization in the last 2 months prior to enrolment or that may require hospitalization (e.g. elective surgery) during the study
* Any clinically significant psychosis or cognitive impairment
* Unlikelihood to comply or complete the study
* Women who are pregnant, lactating or planning to become pregnant during the study period

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-09 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Baseline change in HbA1c at month 3 and 6 between paired testing and control arms for each of the 3 patient segments. | 6 months

SECONDARY OUTCOMES:
Proportion of patients who achieve good glycemic control (HbA1c≤7%) | 6 months

OTHER OUTCOMES:
Baseline change in quality of life score (based on Chinese Normal Audit of Diabetes-Dependent Quality of Life Questionnaire) | 6 months
Baseline change in self-care scores (based on Diabetes Self-Efficacy Scale Questionnaire) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Weiping Jia, MD, PHD, Principal Investigator — Shanghai 6th People's Hospital
Locations (1):
- Weiping Jia, Shanghai, China

REFERENCES:
- [Derived] Shen Y, Zhu W, Lu L, Lu F, Kan K, Bao Y, Zhou J, Jia W. Contribution of structured self-monitoring of blood glucose to self-efficacy in poorly controlled diabetes patients in China. Diabetes Metab Res Rev. 2019 Jan;35(1):e3067. doi: 10.1002/dmrr.3067. Epub 2018 Sep 24. PMID 30144264